CLINICAL TRIAL: NCT00447096
Title: rTMS (Repetitive Transcranial Magnetic Stimulation) for Acute Treatment of Depressed Phase of Bipolar Disorder Type II
Brief Title: rTMS for Treatment of Depressed Phase of Bipolar Disorder Type II
Acronym: rTMS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No results, funding terminated and PI no longer at institution
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Stanley Medical Research Institute (Other); Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102006-040
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Type II; Depression; rTMS
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental): Treatment arm will receive treatment 5 days a week for 6 weeks. Repetitive transcranial magnetic stimulation (rTMS) treatment.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham Arm (Sham Comparator): Sham Arm will not receive any stimulation 5 days a week for 6 weeks. Sham transcranial magnetic stimulation.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Repetitive transcranial magnetic stimulation (rTMS).

SUMMARY:
This research study evaluates an experimental device for the treatment of the depressed phase of Bipolar Disorder Type II. Repetitive Transcranial Magnetic Stimulation (rTMS) is an experimental procedure where a device delivers an alternating magnetic field to a focal area of the brain. When the coil is placed against the scalp on the left frontal area of the head, the magnetic field is focused to a region of the brain that is thought to be involved in depression. This study is intended to test if rTMS can affect this region of the brain in a way that improves the symptoms of depression related to Bipolar Disorder Type II. The purpose of this study is to obtain safety and efficacy information regarding the use of rTMS(Repetitive Transcranial Magnetic Stimulation) for patients in the depressed phase of Bipolar Disorder Type II.

DETAILED DESCRIPTION:
This is a double-blind randomized controlled trial of rTMS for outpatients in the depressive phase of BD-II. Participants will be evaluated at UT Southwestern Medical Center at Dallas. Forty eligible subjects will be randomized to either active treatment (n=20) or sham (no stimulation, n=20). Each subject will receive treatment 5 days per week for a total of 6 weeks. At the end of the 6 weeks, those who remain depressed will have the option of receiving 6 additional weeks of open rTMS treatment. We require these participants to meet the same eligibility criteria in the open phase (i.e. MADRS ≥15, YMRS <12) as in the initial double blind phase. At the completion of treatment, a follow-up appointment will be scheduled with a study physician to ensure that the participant is properly transitioning to clinical care and is not having a significant change in clinical status. Those who do not already have a treating physician will be referred to a new provider.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged 18-55 years old
* Meet DSM-IV criteria for Bipolar Affective Disorder Type II, depressed phase without psychosis as determined by Structured Clinical Interview for DSM-IV
* A MADRS ≥ 15 at Initial Visit, and at Prior to TMS Evaluation
* A Young Mania Rating Scale < 12 at Initial Visit and at Prior to TMS Evaluation
* Duration of current episode of depression >2 months but ≤ 1 year of unsuccessful treatment
* On stable medication and/or psychotherapy for 1 month and clinically appropriate to maintain for duration of trial
* Cognitively intact (Folstein MMSE score >24).
* Clinically competent to give informed written consent

Exclusion Criteria:

* History of epilepsy or seizure disorder, mass brain lesions, cerebrovascular accident, metal in the skull, a history of major head trauma, or any neurologic condition likely to increase risk of rTMS.
* Suicidal risk that precludes safe participation defined as score of 5 or 6 on MADRS item 10 Suicidal Thoughts or clinical impression that the subject is at significant risk for suicide.
* History of any DSM-IV Axis I diagnosis other than Bipolar Affective Disorder Type II, depressed phase, simple phobia and generalized anxiety disorder (GAD) in the last year
* Lifetime history of schizophrenia, schizoaffective, or other psychotic disorder, bipolar disorder type I, dementia, dissociative disorders, and sexual and gender identity disorder
* Personality disorder that makes participation in the trial difficult
* Greater than or equal to 8 episodes of mood disturbance in the previous 12 months
* Greater than 4 unsuccessful treatments in current episode
* History of Substance Abuse or Dependence (DSM-IV) in the last year except nicotine and caffeine
* Positive urine drug test during screening
* Taking any medication that significantly lowers the seizure threshold (e.g. lithium, stimulants, bupropion, TCAs, antipsychotics, theophylline, etc.)
* Unstable medical conditions that precludes safe participation in rTMS treatment trial
* Known or suspected pregnancy
* Women of child-bearing potential not using medically accepted form of contraception when engaged in sexual intercourse
* Any metal or device implants that would increase risk of rTMS
* Unable to determine the motor threshold in the subject
* History of Vagus Nerve Stimulation
* Currently in another investigational study
* Prior electroconvulsive therapy failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
QIDS-C (Quick Inventory of Depressive Symptomatology-Clinical Rated) | 3 year

SECONDARY OUTCOMES:
MADRS(Montgomery Asberg Depression Rating Scale) | 3 year
IDS-C (Inventory of Depressive Symptomatology- Clinician Rated) | 3 year
QIDS-SR (Quick Inventory of Depressive Symptomatology-Self Report) | 3 year
YMRS (Young Mania Rating Scale) | 3 year
Neuropsychological Testing | 3 year
rTMS safety/adverse events | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: F. Andrew Kozel, MD, MSCR, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States